CLINICAL TRIAL: NCT02578966
Title: Impact of Preventive Child Oral Health Programs in Primary Health Care.
Brief Title: Cohort Zero Caries
Acronym: CZC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Daniel Demétrio Faustino da Silva, Dentist, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HNSC-CZC
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries; Early Childhood Caries
Keywords: Early Childhood Caries; Randomized clinical trial; Motivational Interviewing
MeSH Terms: conditions — Dental Caries | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interview (Experimental): INTERVENTION GROUP: in this group, composed of 6 UBS, the children and their respective mothers/fathers/responsible adults will be attended by the dentists at least once a year with an approach based on the Motivational Interview.
  Interventions: Behavioral: Motivational Interview
- Traditional health education (Active Comparator): CONTROL GROUP: in this group, composed of 6 UBS, the children and their respective mother/fathers/responsible adults will be attended by the dentists at least once a year based on the recommendations by the Brazilian Ministry of Health (BRASIL,2008-a) and on SSC-GHC's protocol (BRASIL, 2008-b). Additionally, the professional guidance script and the parents' booklet of SSC-GHC's oral health Program may be used.
  Interventions: Other: Traditional health education

INTERVENTIONS:
Behavioral: Motivational Interview
  Arms: Motivational Interview
Other: Traditional health education
  Arms: Traditional health education

SUMMARY:
The purpose of this study is to compare the effectiveness of a traditional oral health educational program and a program based on the theories of the Motivational Interview directed to the child's mothers/fathers/responsible parents to reduce childhood caries (2 and 3 years of age).

DETAILED DESCRIPTION:
Early Childhood Caries - ECC - is a highly prevalent and severe disease that affects children during their first years of life and, hence, requires early interventions and approaches, on an individual and collective basis. Early childhood is the ideal period to introduce good habits and begin an educational/preventive oral health program; however, family participation is utmost important, especially because the child's parents or responsible adults tend to pass improper knowledge on oral health care in this stage of life. Once prioritizing educational actions directed to this audience in primary health care is essential, Grupo Hospitalar Conceição's (Conceição Hospital Group - GHC) Community Health Service implemented, in its 12 Basic Health Units (UBS), an oral health action program with the goal that all children born after 2010 have at least one dental appointment in their first, second and third year of life. In these appointments, the child's oral health conditions are evaluated and their mother/father or responsible adult receive guidance on proper oral health care; however, little is known on the effectiveness of these preventive programs and what is their impact on ECC reduction in the population. With the purpose of qualifying oral health care strategies at the Brazilian Unified Health System's Primary Health Care (APS-SUS), with a scientific background, it is necessary to assess the effectiveness of these programmatic actions in comparison with conventional dental care by free demand. In light of this, this study has a technological innovation character, with a potential to be directly applicable in the oral health care staff of the Family Health Strategy program throughout Brazil.

The purpose of this study is to compare the effectiveness of a traditional oral health educational program and a program based on the theories of the Motivational Interview directed to the child's mothers/fathers/responsible parents to reduce childhood caries (2 and 3 years of age).

Randomized clinical trial nested in a cohort. The study will be conducted at SSC-GHC, which is composed of 12 Basic Health Units (UBS) located in the Northern region of the city of Porto Alegre, RS-Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Children born in 2014 in the attended territory of 12 Basic Health Units of the Community Health Service of Grupo Hospitalar Conceição, located in the city of Porto Alegre, Rio Grande do Sul, Brazil and who are correctly registered and under follow-up medical attention in the Children Program;
* Mothers/fathers/responsible adults: the person responsible for the child's oral health care and who follows all dental appointments in the health unit will be considered.

Exclusion Criteria:

* Children with special needs or syndromes;
* Children who left the attended territory of Community Health Service of Grupo Hospitalar Conceição health units for more than 6 consecutive months;
* Mothers/fathers/responsible adults without cognitive conditions to answer the study's surveys.

Ages: 12 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 650 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reducing the prevalence of Early Childhood Caries after 3 years of follow verified by the ICDAS index (International Caries Detection & Assessment System) from the realization of reduction of at least 30% of the index pre and post intervention. | three years

REFERENCES:
- [Derived] Colvara BC, Faustino-Silva DD, Meyer E, Hugo FN, Hilgert JB, Celeste RK. Motivational Interviewing in Preventing Early Childhood Caries in Primary Healthcare: A Community-based Randomized Cluster Trial. J Pediatr. 2018 Oct;201:190-195. doi: 10.1016/j.jpeds.2018.05.016. Epub 2018 Jun 6. PMID 29885752